CLINICAL TRIAL: NCT04215471
Title: The Safety and Feasibility of NeoAdjuvant Therapy With Immunoreagent (PD-L1 Antibody SHR-1316) for Resectable Oesophageal Squamous Cell carciNoma (NATION1907II)
Brief Title: NeoAdjuvant Therapy With Immunoreagent (SHR-1316) for Resectable Oesophageal Squamous Cell carciNoma
Acronym: NATION1907II
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: B2019-205R
Record Dates: First submitted 2019-12-27; First posted 2020-01-02 (Actual); Last update posted 2022-06-14 (Actual); Status verified 2022-06

CONDITIONS: Oesophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- NeoAdjuvant Therapy With PD-L1 Antibody SHR-1316 group (Experimental): Patients will receive the neoadjuvant therapy with SHR-1316 followed by the operation.
  Interventions: Drug: PD-L1 Antibody SHR-1316

INTERVENTIONS:
Drug: PD-L1 Antibody SHR-1316 — Neoadjuvant therapy with immunoreagent (PD-L1 antibody SHR-1316) for resectable oesophageal squamous cell carcinoma
  Other Names: PD-L1 antibody

SUMMARY:
The investigators will conduct a prospective, single-arm study to evaluate the safety and feasibility of neoadjuvant therapy with anti-PD-L1 antibody (SHR-1316, Hengrui Medicine) in patients with resectable esophageal squamous cell carcinoma (ESCC).

DETAILED DESCRIPTION:
Host immunity is critical to the development and progression of tumor. PD-1 is the co-inhibitory receptor in many immunity cells while PD-L1, the ligands for PD-1, is expressed in tumor cell and is associated with prognosis. Previous studies have shown that anti-PD-1/PD-L1 antibody had durable responses in patients with advanced malignant tumors such as melanoma, renal cell cancer, lung cancer and esophagus cancer. SHR-1316 (Hengrui Medicine, China), anti-PD-L1 antibody, could induce the elevated secretion of interferon (IFN)-α and showed significant tumor-suppression effect in vivo. The phase III clinical trial on the SHR-1316 versus placebo combines with carboplatin and etoposide in the patients with small cell lung cancer is currently being studied (SHR-1316-III-301).

Esophagus cancer usually has a poor prognosis and esophagus squamous cell carcinoma (ESCC) is the main histological type in China. Combination with operation and neoadjuvant therapy including radiotherapy or/and chemotherapy is considered the standard therapy for local advanced esophagus cancer. However, no studies focused on the neoadjuvant immunotherapy in resectable esophagus have been reported.

Therefore, the investigators will conduct a prospective, single-arm study to evaluate the safety and feasibility of neoadjuvant therapy with anti-PD-L1 antibody (SHR-1316, Hengrui Medicine) in patients with resectable ESCC. The primary objectives included the tumor regression grade, adverse event, safety of operation, complications and 30-day mortality. Our study will also explore the relation of tumor immune milieu, circulating immune cells, soluble factors, circulating tumor cell in the patients. Data from our study will provide the basis for further prospective clinical trials (Phase III). Finally, the investigators aim to discover the biomarkers of response and toxicity to allow patients with ESCC derive more benefit from immunotherapy and minimize the risk of toxicity.

ELIGIBILITY:
Inclusion Criteria:

* The patients should be diagnosed with squamous cell cancer by gastroscopic biopsies and the tissue samples should be collected before the treatment.
* The primary tumor should be located in the thorax; the primary site is decided by the upper margin of the mass (upper thoracic esophagus: from the thoracic inlet to inferior margin of azygos arch, the endoscopic examination shows 20-25cm to the incisor; middle thoracic esophagus: from inferior margin of azygos arch to the inferior pulmonary vein level, the endoscopic examination shows 25-30cm to the incisor; lower thoracic esophagus: from the inferior pulmonary vein level to the stomach, the endoscopic examination shows 30-40cm to the incisor).
* The patients should be evaluated to be able to have surgical resection before the surgery according to the examinations (use enhanced thoracic and abdominal CT, cervical lymph node ultrasound to evaluate whether the tumor has obvious invasion, whether there are enlarged mediastinal lymph nodes; use examinations including positron emission computed tomography (PET-CT), endoscopic ultrasonography (EUS) to make further clinical staging if considering the primary tumor as T4b, multiple mediastinal lymph nodes metastasis or distant metastasis).
* The patients should be at the range of 18-75 years old, Eastern Cooperative Oncology Group (ECOG) 0-1, the estimated survival time should be over 12 months.
* The recipients should have no functional disorders in main organs. Blood routines, functions of lung, liver, kidney and heart should be basically normal, the label test index should accord with the demands as follows: Blood: white blood cell count (WBC)>4.0*10^9/L, absolute neutrophil count (ANC)≥2.0*10^9/L, platelet count (PLT)>100*10^9/L, hemoglobin (HBG)>90g/L; Pulmonary function: Forced Expiratory Volume in the first second (FEV1)≥1.2 L, FEV1%≥50%, carbon monoxide diffusing capacity (DLCO)≥50%; Liver function: Serum bilirubin should be lower than 1.5 times of the maximum normal value; Alanine aminotransferase (ALT) and Aspartate transaminase (AST) should be lower than 1.5 times of the maximum normal value; Renal function: serum creatinine (SCr)≤120μmol/L creatinine clearance rate （CCr）≥60ml/min;
* The patients should be able to understand our research and sign the informed consent.

Exclusion Criteria:

Exclusion criteria related to cancer:

* The stage of tumor is T4b (AJCC/International Union Against Cancer (UICC) 8th Edition) which can not be resected according to imaging examinations like thoracic and abdominal enhanced CT, cervical lymph nodes ultrasound, whole body PET-CT scan (optional) or endobronchial ultrasonography (EBUS) (optional); several enlarged lymph nodes existed (≥3 estimated lymph nodes metastasis); multiple station enlarged lymph nodes existed (≥2 estimated stations of lymph nodes metastasis); distant metastasis existed.
* The patients have accepted or are on the process of other chemotherapy, radiotherapy or targeted therapy.
* Endoscopic examination shows non-squamous carcinoma.
* The patients have history of other tumors (not include history of carcinoma in situ of the cervix, cured localized skin basal cell carcinoma).

Other exclusion criteria:

* The patients have history of autoimmune diseases.
* The patients have recently taken steroids or immune immunosuppressive agents or are taking them.
* The patients have history of immunotherapy.
* The patients have history of severe hypersensitivity to antibody drugs.
* The patients have history of chronic or recurrent autoimmune diseases.
* The patients have interstitial lung disease, pulmonary fibrosis, diverticulitis or systematic ulcerative gastritis.
* The patients have proved history of congestive heart failure, angina without good control with medicine; ECG-proved penetrating myocardial infarction; hypertension with bad control; valvulopathy with clinical significance; arrhythmia with high risk and out of control.
* The patients have severe systematic intercurrent disease, such as active infection or poorly controlled diabetes; coagulation disorders; hemorrhagic tendency or under treatment of thrombolysis or anticoagulant therapy.
* Female who is positive for serum pregnancy test or during lactation period, or people at child bearing stage who are reluctant to use contraception measures during the research.
* The patients have active infection of HIV, hepatitis B virus (HBV), hepatitis C virus (HCV) or be HIV serum positive; or HBV, HCV RNA positive.
* The patients are allergic for any of the drugs in the research.
* The patients have history of organ transplantation (including autologous bone marrow transplantation and peripheral stem cell transplantation.
* The patients have history of peripheral nerve system disorders, obvious mental disorders or central nerve system disorders.
* The patients are using other anti-tumor drugs.
* The patients attend other clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-07-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response | Through the study completion, an average of 12 weeks
  The primary endpoint is objective response (according to the Response Evaluation Criteria In Solid Tumors, version 1.1).

SECONDARY OUTCOMES:
Adverse events and treatment-related adverse events | Through the study completion, an average of 12 weeks
  Number of participants with treatment-related adverse events as assessed by CTCAE v4.0
Correlation between genetic profile and tumor response | Through the study completion, an average of 12 weeks
  Genetic profile (assessed by whole exome sequencing, T-cell receptor sequencing, RNA sequencing) will be correlated with tumor objective response

CONTACTS AND LOCATIONS:
Overall Officials: Lijie Tan, MD, PhD, Principal Investigator — Shanghai Zhongshan Hospital
Locations (1):
- 180 Fenglin Road, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data (IPD) will be shared
Supporting Information: Study Protocol
Time Frame: After the study is completed.
Access Criteria: IPD will be uploaded for access of other researchers.

REFERENCES:
- [Derived] Yin J, Yuan J, Li Y, Fang Y, Wang R, Jiao H, Tang H, Zhang S, Lin S, Su F, Gu J, Jiang T, Lin D, Huang Z, Du C, Wu K, Tan L, Zhou Q. Neoadjuvant adebrelimab in locally advanced resectable esophageal squamous cell carcinoma: a phase 1b trial. Nat Med. 2023 Aug;29(8):2068-2078. doi: 10.1038/s41591-023-02469-3. Epub 2023 Jul 24. PMID 37488287